CLINICAL TRIAL: NCT07000214
Title: Peripheral Magnetic Stimulation With Balance Training to Decrease Fall Risks in Older Patients With Diabetic Polyneuropathy
Brief Title: Peripheral Magnetic Stimulation With Balance Training to Decrease Fall Risks in Diabetic Polyneuropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Komwudh Konchalard, Physiatrist, Department of Rehabilitation Medicine, Queen Savang Vadhana Memorial Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010/2568
Record Dates: First submitted 2025-05-29; First posted 2025-06-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Polyneuropathy
Keywords: diabetic polyneuropathy; fall risk; peripheral magnetic stimulation; balance training
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peripheral magnetic stimulation with balance training (rPMS-BT) (Experimental): The participants will undergo a warm-up exercise involving ankle dorsiflexion, with concurrent rPMS applied to the tibialis anterior of each leg. Following the warm-up, participants will stand on the MAGBATA platform and perform one-leg stance exercises while rPMS is applied to the plantar surface of the foot. This procedure will be repeated for the other leg.
  Interventions: Device: Peripheral magnetic stimulation; Behavioral: Balance training
- Sham stimulation with balance training (Sham-BT) (Sham Comparator): The sham comparator group will receive the same procedure as the interventional group, but with sham stimulation during both the warm-up and one-leg stance exercise.
  Interventions: Behavioral: Balance training; Other: Sham stimulation

INTERVENTIONS:
Device: Peripheral magnetic stimulation — During the warm-up exercise, 10-Hz rPMS will be applied to the tibialis anterior with an on-time of 4 seconds (40 pulses per train), followed by an off-time (inter-train interval) of 8 seconds, for a total of 25 trains for each leg. During the one-leg stance exercise, 20-Hz rPMS will be applied to the plantar surface of the standing foot for 3 seconds of on-time (60 pulses per train), followed by 12 seconds of off-time, for a total of 20 trains for each foot. Stimulation intensity will be set at 110% of MCT for the warm-up exercise and 120% of MCT for the treatment during the one-leg stance exercise.
  Arms: Peripheral magnetic stimulation with balance training (rPMS-BT)
Behavioral: Balance training — The warm-up exercise consists of 25 repetitions of 4-second active contractions of the tibialis anterior muscle in each leg while seated. Following the warm-up, participants will stand on the MAGBATA platform and perform 20 cycles of one-leg stance exercises under the supervision of a physiotherapist. Each cycle lasts 20 seconds, consisting of 3 seconds of one-leg stance while the other leg is raised about 10 centimeters above the ground, followed by 12 seconds of rest during which the participant stands on both legs, keeping their arms close to their body and hands free. The same sequence will then be repeated for the other leg. To prevent falling, participants will wear a safety belt around the waist, allowing the physiotherapist to assist if they lose balance. Participants will also be allowed to grab the walker positioned in front of them to prevent falling.
Other: Sham stimulation — During the warm-up exercise, the stimulation coil will be placed perpendicular to the participants' shin. The same parameter settings will be used, except for the intensity, which will be set at 30% of the maximum stimulator output (MSO). Sham stimulation during the one-leg stance exercise is achieved by disconnecting the coil mounted in MAGBATA and placing an alternate coil, connected to the magnetic stimulator placed behind the participants so they can hear a clicking pattern similar to that of the rPMS-BT arm.
  Arms: Sham stimulation with balance training (Sham-BT)

SUMMARY:
This study aims to determine whether peripheral magnetic stimulation (PMS) during balance training in patients with diabetic polyneuropathy reduces fall risk, as measured by balance tests, and lessens disease severity compared to balance training with sham stimulation.

This proof-of-concept study will utilize the Magnetic and Balance Training Activator (MAGBATA), a platform mounted with a magnetic stimulation coil that delivers electromagnetic pulses directly to the plantar surfaces of the feet while patients stand. A racetrack coil (RT-120), connected to the MagPro X100 magnetic stimulator with MagOption (MagVenture, Farum, Denmark), will be used. Parameters for the repetitive peripheral magnetic stimulation (rPMS) protocol will be configured to facilitate sensory input, enhance brain plasticity, and promote axonal regeneration.

DETAILED DESCRIPTION:
This single-center randomized controlled trial will use a two-group parallel design and include 40 patients with diabetic polyneuropathy who meet the eligibility criteria. Participants will be randomly assigned to either the active intervention group or the control group.

The active intervention group will receive a warm-up exercise consisting of 25 repetitions of ankle dorsiflexion with concurrent 10 Hz rPMS applied to the tibialis anterior of each leg. Following the warm-up, participants will stand on the MAGBATA platform and perform 20 cycles of one-leg stance exercises under the supervision of a physiotherapist. Each cycle lasts 20 seconds and consists of 3 seconds of 20 Hz rPMS applied to the plantar surface of the foot while the participant stands on one leg, followed by 12 seconds of rest during which the participant stands on both legs. The same sequence will then be repeated for the other leg. Stimulation intensity will be determined prior to the warm-up. The coil will be placed over the tibialis anterior to determine the minimal contraction threshold (MCT), defined as the lowest intensity that produces a visible contraction. The stimulation intensity will be set at 110% of the MCT for the warm-up exercise and 120% for the treatment during balance exercises.

The control group will receive the same procedure, but with sham stimulation during both the warm-up and one-leg stance phases.

The intervention will consist of 8 sessions, conducted twice per week with at least one day of rest between sessions. Outcome assessments include one-leg stance test (OLST) with eyes open, timed up and go test (TUGT), and short physical performance battery (SPPB); these assessments will be conducted at baseline and after the 4-week intervention. Additionally, a rehabilitation physician, blinded to group allocation, will perform electrophysiologic studies at baseline and week 8 to assess disease severity. These studies will include bilateral measurements of sural nerve amplitude and conduction velocity, tibial compound motor action potential (CMAP) amplitude and conduction velocity, and tibial F-wave latency.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 with any symptoms of distal polyneuropathy, including numbness, paresthesia, dysesthesia, or lower leg weakness.
* Abnormal 10g monofilament test.
* Abnormal one-leg stance test (OLST) with eyes open.

Exclusion Criteria:

* Chronic foot ulceration.
* Severe leg or foot pain not controllable with medications or other interventions.
* Significant foot deformity, including severe pes cavus, severe claw toe, or toe amputation.
* Body mass index (BMI) over 30 kg/m².
* Visual acuity less than 20/100 after correction with glasses or contact lenses.
* Postural instability or coordination disorders resulting from musculoskeletal, vestibular, or central nervous system conditions.
* Symptoms such as confusion, drowsiness, dizziness, or a high risk of falls due to any disease or recent medication changes within a two-week period.
* Presence of cardiac pacemaker, knee prosthesis, or metal implants in the lower legs.
* Inability to walk or stand for at least 5 minutes.
* Inability to understand, comprehend, or follow instructions required to conduct the study, or to provide informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
One-leg standing balance test (OLST) | From enrollment to the end of treatment (week 4).
  Participants stand on the floor with their eyes open and arms relaxed at the sides of the body. They are instructed to lift the opposite foot off the floor, flex the knee to 90 degrees, and position the lifted foot behind the body, maintaining balance on the tested leg for as long as possible. The assessor begins timing when the participant's foot leaves the floor and stops timing if the participant sways, extends either arm to maintain balance, or successfully holds the position for 30 seconds. The test is then repeated on the opposite leg. The durations from both legs are summed and reported in seconds.

SECONDARY OUTCOMES:
Timed up and go test (TUGT) | From enrollment to the end of treatment (week 4).
  Participants sit on a chair with a seat height between 44 and 47 cm, with their back resting against the backrest. The assessor instructs them to walk to a marked point 3 meters straight ahead and then return to sit on the chair. Timing begins when the participant's back leaves the backrest and stops when they return to the chair and their back touches the backrest. The test is performed twice, and the best performance with shorter duration in seconds, will be recorded.
Short physical performance battery (SPPB) | From enrollment to the end of treatment (week 4).
  The Short Physical Performance Battery (SPPB) includes three subtests: gait speed, chair stand, and balance. Each test scored from 0 to 4and are summed up to give a total score ranging from 0 to 12.
  Gait speed: Participants are instructed to walk at their normal pace over a distance of 4 meters. The assessor times each trial from the start of walking until the participant reaches the end.
  Chair stand test: Participants are instructed to rise from a seated position to standing five times, keeping their arms crossed at chest level. The assessor starts timing when the participant's buttocks leave the chair and stops when they return to the seat after the fifth stand.
  Balance test on both feet: Participants first stand with feet together for 10 seconds to earn 1 point, then in semi-tandem with the heel beside the mid-foot for 10 seconds to earn another point, and finally in full tandem for 10 seconds to earn 2 points.
Severity grading based on nerve conduction velocity | From enrollment to week 8.
  Nerve conduction study will be performed using the electrodiagnostic unit, Sierra Summit (Cadwell, Kennewick, WA, USA). Bilateral sural and tibial nerves will be tested, measuring parameters including conduction velocity, sensory nerve action potential (SNAP) amplitude of the sural nerves, compound motor action potential (CMAP) amplitudes of the tibial nerves, F-wave latency of the tibial nerves, and the presence of A-waves. Severity will be classified into five categories, from grade 0 to 4, with higher grades indicating greater severity, based on the algorithm for grading diabetic polyneuropathy by Baba classification. The outcome will be categorized as 'improved' if the grade at week 8 is lower than at baseline, and 'not improved' if the grade at week 8 remains unchanged or increases.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data related to the primary and secondary outcomes of all participants will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication; for 2 years.
Access Criteria: IPD will be shared upon reasonable request by email with researchers conducting similar studies or performing meta-analyses. The process will require approval by the Institutional Review Board (IRB) and may also require a data use agreement.

REFERENCES:
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Himeno T, Kamiya H, Nakamura J. Lumos for the long trail: Strategies for clinical diagnosis and severity staging for diabetic polyneuropathy and future directions. J Diabetes Investig. 2020 Jan;11(1):5-16. doi: 10.1111/jdi.13173. Epub 2019 Dec 1. PMID 31677343
- [Background] Xu S, Ito A, Zhao Z, Nakahara R, Tai C, Miyamoto F, Kuroki H, Aoyama T. Repetitive magnetic stimulation prevents dorsal root ganglion neuron death and enhances nerve regeneration in a sciatic nerve injury rat model. Sci Rep. 2024 Aug 16;14(1):19016. doi: 10.1038/s41598-024-69251-4. PMID 39152157
- [Background] Yan T, Liang M, Peng J, Yu Q, Li Y, Yang J, Zhang S, Wang C. Cortical Mechanisms Underlying Effects of Repetitive Peripheral Magnetic Stimulation on Dynamic and Static Postural Control in Patients with Chronic Non-Specific Low Back Pain: A Double-Blind Randomized Clinical Trial. Pain Ther. 2024 Aug;13(4):953-970. doi: 10.1007/s40122-024-00613-6. Epub 2024 Jun 19. PMID 38896200
- [Background] Alissa N, Shipper AG, Zilliox L, Westlake KP. A Systematic Review of the Effect of Physical Rehabilitation on Balance in People with Diabetic Peripheral Neuropathy Who are at Risk of Falling. Clin Interv Aging. 2024 Jul 19;19:1325-1339. doi: 10.2147/CIA.S459492. eCollection 2024. PMID 39050517
- [Background] Baek J, Park N, Lee B, Jee S, Yang S, Kang S. Effects of Repetitive Peripheral Magnetic Stimulation Over Vastus Lateralis in Patients After Hip Replacement Surgery. Ann Rehabil Med. 2018 Feb;42(1):67-75. doi: 10.5535/arm.2018.42.1.67. Epub 2018 Feb 28. PMID 29560326
- [Background] Smith S, Ravikumar R, Carvalho C, Normahani P, Lane T, Davies AH. Neuromuscular electrical stimulation for the treatment of diabetic sensorimotor polyneuropathy: A prospective, cohort, proof-of-concept study. Neurophysiol Clin. 2024 May;54(3):102943. doi: 10.1016/j.neucli.2024.102943. Epub 2024 Feb 29. PMID 38422719
- [Background] Ahmad I, Noohu MM, Verma S, Singla D, Hussain ME. Effect of sensorimotor training on balance measures and proprioception among middle and older age adults with diabetic peripheral neuropathy. Gait Posture. 2019 Oct;74:114-120. doi: 10.1016/j.gaitpost.2019.08.018. Epub 2019 Aug 30. PMID 31499405
- [Background] Dana E, Tran C, Osokin E, Westwood D, Moayedi M, Sabhaya P, Khan JS. Peripheral magnetic stimulation for chronic peripheral neuropathic pain: A systematic review and meta-analysis. Pain Pract. 2024 Apr;24(4):647-658. doi: 10.1111/papr.13332. Epub 2023 Dec 16. PMID 38102884